CLINICAL TRIAL: NCT06879587
Title: Assessing the Safety and Effectiveness of Bacillus Coagulans BC99 in Relieving Functional Constipation in Adults Based on Randomized, Double-Blind, Placebo-Controlled Trials
Brief Title: Probiotics Alleviate Functional Constipation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024019
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Participants receive one sachet per day containing probiotic BC99 and maltodextrin (Week 0 to Week8).
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): Participants receive one sachet per day containing maltodextrin only, serving as the placebo(Week 0 to Week8).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — During the intervention, participants could take BC99 daily and record any adverse reactions. Participants filled out questionnaires and collected stool and serum samples, which were used to detect and analyze the improvement of participants' constipation function.
  Arms: Probiotic Group
Dietary Supplement: Placebo — During the intervention, participants could take maltodextrin daily and record any adverse reactions. Participants filled out questionnaires and collected stool and serum samples, which were used to detect and analyze the improvement of participants' constipation function.
  Arms: Placebo Group

SUMMARY:
To investigate the clinical effects of probiotics in relieving chronic constipation in adults, and evaluate the improvement of symptoms in patients with constipation as well as their impacts on gastrointestinal function, immunity, and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults aged 18-70 who meet the following Rome-IV diagnostic criteria for Functional constipation:

   i. If the following symptoms started at least 6 months ago and have been present for the past 3 months with two or more of the following:
   1. Straining during more than 25% of defecations
   2. Lumpy or hard stools (Bristol Stool Form Scale 1-2) more than 25% of defecations
   3. Sensation of incomplete evacuation more than 25% of defecations
   4. Sensation of anorectal obstruction/blockage more than 25% of defecations
   5. Manual maneuvers to facilitate more than 25% of defecations (e.g., digital evacuation, support of the pelvic floor)
   6. Fewer than three SBM per week ii Loose stools are rarely present without the use of laxatives iii. Insufficient criteria for irritable bowel syndrome.
2. Able to complete the study according to the requirements of the trial protocol;
3. Patients who have signed the informed consent form;
4. Research participants (including male participants) who have no fertility plans from 14 days before screening until 6 months after the end of the trial and are willing to take effective contraceptive measures.

Only those who meet all the above conditions can be selected for the study. -

Exclusion Criteria:

1. The use of probiotics, prebiotics, or antibiotics within 2 weeks of enrollment.
2. Regular use of a high-fiber diet, as measured by the recommended food score (RFS);
3. Regular use of medications affecting bowel habits, such as irritable bowel syndrome, functional bloating, and functional diarrhea.
4. Currently have, or have had in the past 2 years, any gastrointestinal conditions such as: Crohn's disease, celiac disease, Ulcerative colitis, Malignant tumor of the colon.
5. Medical history of cardiovascular, liver, or renal diseases; alcoholics.
6. Hypersensitivity to probiotics or the ingredients used in this study.
7. Pregnancy or breastfeeding.
8. Participation in another clinical trial in the 3 months before enrollment. All participants provided written informed consent. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-09-08 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Change in colonic transit time (CTT) from baseline to 8 weeks | Week 0 and Week 8
  Colonic transit time (hours) was measured by radiolabmarking, and the reduction from baseline was an indicator of effectiveness.
Change in Patient Assessment of Constipation Symptoms (PAC-SYM) score from baseline to 8 weeks. | Week 0 and Week 8
  The PAC-SYM questionnaire was used to assess the severity of constipation symptoms (12 items, 0-4 Likert score), with a total score ranging from 0-48 (the lower the score, the milder the symptoms). The magnitude of the decline from the baseline score is an indicator of effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Technology, Zhengzhou, Henan, China